CLINICAL TRIAL: NCT00868959
Title: A 24-Week, Flexible-Dose, Open-Label Extension Study of Lurasidone for the Treatment of Bipolar I Depression
Brief Title: Lurasidone - A 24-week Extension Study of Patients With Bipolar I Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1050256; EUDRACT No. 2008-007483-42
Record Dates: First submitted 2009-03-23; First posted 2009-03-25 (Estimated); Results first posted 2014-04-01 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-03

CONDITIONS: Bipolar Depression
Keywords: Bipolar; Depression; Lurasidone; Latuda
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lurasidone (Experimental)
  Interventions: Drug: lurasidone

INTERVENTIONS:
Drug: lurasidone — Lurasidone 20-120 mg/d Flexibly Dosed - 24 weeks

SUMMARY:
This clinical study is designed to test the hypothesis that lurasidone is effective, tolerable, and safe for the treatment of patients with bipolar I depression

ELIGIBILITY:
Inclusion Criteria:

* Subject is judged by the investigator to be suitable for participation in a 24-week clinical trial involving open-label lurasidone treatment
* Subject has completed the 6-week treatment period and all required assessments on the final study visit (Day 42, Visit 8) of either Study D1050235, NCT#00868452 or Study D1050236, NCT#008668699.

Exclusion Criteria:

* Imminent risk of suicide, injury to self or to others, or damage to property
* Subject has evidence of severe movement disorders.
* Subject tests positive for drugs of abuse (at Visit 8 in Study D1050235, NCT#00868452 or D1050236, NCT#008688699).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 817 (Actual)
Dates: Start 2009-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (151):
- United States (58):
  - Woodland International Research Inc, Little Rock, Arkansas
  - South Coast Clinical Trials Inc., Anaheim, California
  - Catalina Research Institute, Chino, California
  - Clinical Innovations Inc., Costa Mesa, California
  - Synergy Escondido, Escondido, California
  - Collaborative Neuroscience Network Inc, Garden Grove, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Florida Clinical Research Center LLC, Maitland, California
  - Excell Research, Inc, Oceanside, California
  - University of California at Irvine Medical Center, Orange, California
  - CNRI - Los Angeles LLC, Pico Rivera, California
  - Clinical Innovations Inc., Riverside, California
  - California Neuropsychopharmacology Clinical Research Instit, San Diego, California
  - Artemis Institute for Clinical Research LLC, San Diego, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - Clinical Innovations Inc., Santa Ana, California
  - Stanford University School of Medicine, Stanford, California
  - Collaborative Neuroscience Network Inc., Torrance, California
  - University of Colorado, Aurora, Colorado
  - MCB Clinical Research Centers-Colorado Springs, Colorado Springs, Colorado
  - Florida Clinical Research Center LLC, Bradenton, Florida
  - Florida Clinical Research Center LLC, Fruitland Park, Florida
  - Accurate Clinical Trials, Kissimmee, Florida
  - Clinical Neuroscience Solutions INc., Orlando, Florida
  - University of South Florida Institute - Tampa, Tampa, Florida
  - Janus Center for Psychiatric Research, West Palm Beach, Florida
  - Northwest Behavioral Research Center, Rosewekk, Georgia
  - Institute for Behavioral Medicine LLC, Smyrna, Georgia
  - American Medical Research, Oak Brook, Illinois
  - Lake Charles Clinical Trials LLC, Lake Charles, Louisiana
  - Booker, J. Gary, MD. APMC, Shreveport, Louisiana
  - Sheppard Pratt Health System, Baltimore, Maryland
  - Capitol Clinical Research, Rockville, Maryland
  - Precise Research Centers, Flowood, Mississippi
  - Midwest Research Group, Saint Charles, Missouri
  - CRI Worldwide, LLC, Willingboro, New Jersey
  - Albuquerque Neuroscience Inc., Albuquerque, New Mexico
  - Social Psychiatry Research Institute, Brooklyn, New York
  - Neurobehavioral Research, Inc, Cedarhurst, New York
  - Village Clinical Research Inc., New York, New York
  - Medical & Behavioral Health Research PC, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Zarzar Psychiatric Associates PLLC, Raleigh, North Carolina
  - Richard H. Weisler & Associates, Raleigh, North Carolina
  - Quest Therapeutics, Avon Lake, Ohio
  - Psychiatric Professional Services Inc, Cincinnati, Ohio
  - Mood Disorders Program-UHCMC, Cleveland, Ohio
  - MetroHealth System, Cleveland, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Summit Research Network (Oregon) Inc., Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Clinical Neuroscience Solutions Inc., Memphis, Tennessee
  - FutureSearch Clinical Trials LP, Austin, Texas
  - FutureSearch Trials, Dallas, Texas
  - Pillar Clinical Research LLC, Dallas, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Wharton Research Center, Wharton, Texas
  - Summit Research Network (Seattle) LLC, Seattle, Washington
- Canada (4):
  - Clinical Research Group Edmonton, Edmonton, Alberta
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - Pierre-Janet Hospital, Gatineau, Quebec
  - Hopital Louis-H Lafontaine, Montreal, Quebec
- Colombia (4):
  - Centro de Investigaciones y Proyectos en Neurociencias CIPNA Investigations, Barranquilla
  - E.S.E. Hospital Mental de Antioquia, Bello
  - Centro de Investigacion y Atencion para la Salud Mental, Bogotá
  - Centro de Investigaciones del Sistema Nerviosa Limitada-Gr, Bogotá
- Czechia (7):
  - Saint Anne, s.r.o., Psychiatricke oddeleni, Brno - Mesto
  - BIALBI s.r.o. Psychiatricke oddeleni, Litoměřice
  - Psychiatricka ambulance Prosek, Lovosicka
  - Vojenska nemocnice Olomouc, Olomouc
  - Clintrial, s.r.o., Prague
  - Psychiatry Trial s.r.o., Prague
  - Medical Services Prague s.r.o., Prague
- France (2):
  - Hopital Caremeau, Service de Psychiatrie A, Nîmes
  - Zans Ritter, Marcel, Orvault
- India (21):
  - S V Medical College, Tirupati, Andh Prad
  - Vijayawada Institute of Mental Health and Neurosciences, Psychiatry, Vijaywada, Andh Prad
  - Brain Mind Behaviour Neurosciences Research Institute, Visakhapatnam, Andh Prad
  - Seth K M School of P G Medicine & Research, Ahmedabad, Gujarat
  - Mental Illness Treatment Rehabilitation Foundation (MITR), Ahmedabad, Gujarat
  - Brij Psychiatry Hospital & Muskaan Research Centre, Vadodara, Gujarat
  - Spandana Nursing Home, Bangalore, Karna
  - Abhava Hospital, Bangalore, Karna
  - K.S. Hegde Medical Academy, Mangalore, Karna
  - Shanti Nursing Home, Aurangabad, Mahara
  - Poona Hospital & Research Center, Pune, Mahara
  - Mahatma Gandhi Institute of Medical Sciences, Wardha, Mahara
  - Cosmos Hospitals-Delhi Psychiatry Center-Dept. of Psychiatry, Delhi, National Capital Territory of Delhi
  - Dr. Tambi's Neuropsychiatry Center, Jaipur, Rajaasthan
  - R.K. Yadav Memorial Mental Health & De-Addiction Hospital Psychiatry, Jaipur, Rajasthan
  - Mahendru Psychiatric Centre, Kanpur, Uttar Prad
  - Manobal Med. Research Centre, Lucknow, Uttar Prad
  - Shree Hatkesh Health Foundation, Gujarat
  - Samvedna Hospitals, Gujarat
  - Chhatrapati Shahuji Maharaj, Lucknow
  - Sujata Dirla Hospital & Research Centre, Mahara
- Japan (6):
  - Ongata Hospital, Hachioji-shi
  - Kohnodai Hp., National Center for Global Health and Medicine, Ichikawa-sha
  - NHO Hizen Psychiatric Center, Kanzaki-gun
  - National Center of Neurology and Psychiatry, Kodaira-shi
  - Asakayama General Hospital, Sakaishi
  - Osaka Institute of Clinical Psychiatry Shin-abuyama Hospital, Takatsuki-shi
- Lithuania (5):
  - Neuromeda, JSC, Kaunas
  - Kaunas Hospital Division Marui Hospital, Public Institution, Kaunas
  - Silutes Mental Health and Psychotherapy Center, JSC, Šilutė
  - Seskines Outpatient Clinic, Public Institution, Vilnius
  - Zirmunai Mental Health Center, Public Institution, Vilnius
- Peru (3):
  - Hospital Nacional Hipolito Unanue, Lima
  - Hospital Nacional Arzobispo Loayza, Lima
  - Clinica Vesalio, Lima
- Poland (2):
  - ZOZ Poradnia Zdrowia Psychicznego, Chełmno
  - Praktyka Lekarska Sensorium S.M.O., Skorzewo
- Romania (6):
  - Spitalul Clinic de Urgenta Militar Central, Bucharest
  - Spitalul Clinic de Psihaiatrie Prof. Dr. Alexandru Obregia, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj, Cluj-Napoca
  - Spitalul Clinic de Neuropsihiatrie Craiova, Craiova
  - Centrul de Recuperare si Reabilitare Gura Ocnitei, Gura Ocniței
  - Spitalul Clinic de Neurologie si Psihiatrie Oradea, Oradea
- Russia (6):
  - Russian State Medical University of RosZdrav, Moscow
  - Moscow Medical Academy name I.M. Sechenov, Moscow
  - City Psychiatric Hospital #2 of St. Nikolay Chudotvorets, Saint Petersburg
  - Bekhterev Scientific Research Psychoneurological Institute, Saint Petersburg
  - Psychoneurology Dispensary #4, Saint Petersburg
  - LLC International Medical Centre "SOGAZ", Saint Petersburg
- Slovakia (8):
  - Nemocnica s poliklinikou Prievidza so sidlom v Bojniciach Psychiatricke oddelenie, Bojnice
  - Psychiatricka ambulancia Mentum, s.r.o., Bratislava
  - Univerzitna nemocnica Bratislava, Nemocnica Ruzinov Psychiatricka klinika, Bratislava
  - Nemocnica s poliklinikou Liptovsky Mikulas Psychiatricke oddelenie, Liptovský Mikuláš
  - PsychoLine s.r.o. Psychiatricka ambulancia, Rimavská Sobota
  - Nemocnica s poliklinikou sv Barbory Roznava a.s. Psychiatricke oddelenie, Rožňava
  - Centrum zdravia R. B.K. s.r.o. Psychiatricka ambulancia, Svidník
  - Pro mente sana s.r.o. Psychiaricka ambulancia, Trenčín
- South Africa (6):
  - Groote Schuur Hospital, Cape Town
  - Cape Trial Centre, Cape Town, W. Cape
  - Paarl Medical Centre, Paarl, W. Cape
  - Clinika, Murray and Roberts Building, Port Elizabeth
  - Dey Clinic, Pretoria, Gauteng
  - Vereeniging Medi-Clinic, Vereeniging, Free State
- Ukraine (13):
  - Regional Clinical Hospital n.a.l.l., Dnipropetrovsk
  - Com. Inst. "Dnipropetrovsk Reg. Cl. Psych. Hosp." DSMA, Dnipropetrovsk
  - Reg. Clin. Psychiatric Hosp. DSMU n.af.M.Gorkiy, Donetsk
  - St.In."Inst. of Neurol., Psych. and Narcol. of the AMSU", Kharkiv
  - Kherson Regional Psychiatric Hospital, Kherson
  - Kyiv City Psychoneurological Hospital #2, Kviv
  - Lviv Reg.St.Cl.Psych.Hosp.Dept.#20, LNMU n.a.D. Halytskiy Chair of Psychiatry, Psychology and Sexololgy, Lviv
  - Odesa SMU, based on Odessa Reg. Psychiatric Hosp.#1, Odesa
  - Reg. Ci.Ps.H.n.a.O.F.Maltsev, Fem.Ac.Gen.Ps. D.5B,HESIU UM, Poltava
  - Crimean republican Clinical Psychiatric Hospital, Simferopol
  - Ternopil Regional Municipal Dispensary, Narcology Dept., Ch. of Neurol. Psych. Narcol. & Med. Psychol., Ternopil
  - Reg. Psych. Hosp.n.a. O.Yuschenko, Dept. #121 VNMI, Vinnitsia
  - Zapor Reg. Cl. Hosp., Zaporizhzhia SMU, ENT Dept., Zaporizhzhia

REFERENCES:
- [Derived] Forester BP, Sajatovic M, Tsai J, Pikalov A, Cucchiaro J, Loebel A. Safety and Effectiveness of Long-Term Treatment with Lurasidone in Older Adults with Bipolar Depression: Post-Hoc Analysis of a 6-Month, Open-Label Study. Am J Geriatr Psychiatry. 2018 Feb;26(2):150-159. doi: 10.1016/j.jagp.2017.08.013. Epub 2017 Oct 10. PMID 29146409

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 817 represents the total number of subjects who provided informed consent and enrolled, which is different from the total number of subjects who were treated with study drug, which was 813.
Period: Overall Study
Arm/Group | Lurasidone
Started | 817 (817 represents total number of subjects who provided informed consent.)
Completed | 559
Not Completed | 258

BASELINE CHARACTERISTICS:
Population: Safety population - received at least one dose of study medication
Arm/Group | Lurasidone
Number analyzed (Participants) | 813
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (12.03)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 790
  >=65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 427
  Male | 386
Region of Enrollment [Number; unit: participants]
  United States | 283
  Slovakia | 19
  Ukraine | 78
  Lithuania | 16
  Russian Federation | 31
  Colombia | 15
  India | 128
  France | 23
  Czech Republic | 108
  Canada | 14
  Poland | 12
  Romania | 9
  Peru | 12
  South Africa | 56
  Japan | 6
  Germany | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious and Non-serious Treatment-emergent Adverse Events Who Have Completed 24 Weeks of Extension Study Treatment
Description: Rate of treatment-emergent adverse events in subjects who have completed (ie, reached 6-week endpoint) of Study D1050235 (NCT00868452), Study D1050236 (NCT00868699) or Study D1050292 (NCT01284517)
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Lurasidone
Number analyzed (Participants) | 813
participants | 529

2. Secondary Outcome: Change From Open-label Extension Baseline to Week 24 (Month 6/LOCF Endpoint) in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a clinician-rated assessment of the subject's level of depression. Ten items are rated on a Likert scale, from 0="Normal" to 6="Most Severe". The MADRS total score is calculated as the sum of ten items: reported sadness, apparent sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. The MADRS total score ranges from 0 to 60. Higher scores are associated with greater severity.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone
Number analyzed (Participants) | 813
units on a scale | -4.4 (10.60)

3. Secondary Outcome: Change From Open-label Extension Baseline to Week 24 (Month 6/LOCF Endpoint) in Clinical Global Impressions Bipolar Version, Severity of Illness (CGI-BP-S) Score (Depression)
Description: This CGI-BP-S is a clinician-rated assessment of the subjects current severity of depression and ranges from 1="Normal, not ill" to 7="Very severly ill". Higher scores are associated with greater severity.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone
Number analyzed (Participants) | 813
units on a scale | -0.58 (1.325)

ADVERSE EVENTS:
Time Frame: 24 Weeks
Description: January 22, 2009 - February 19, 2013 - recruitment period
Arm/Group | Lurasidone
Serious Adverse Events (participants affected / at risk) | 24/813
Other Adverse Events (participants affected / at risk) | 246/813
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone (N=813)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Disease Progression (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Hand Fracture (Injury, poisoning and procedural complications) | 1 (1)
Humerous Fracture (Injury, poisoning and procedural complications) | 1 (1)
Radius Fracture (Injury, poisoning and procedural complications) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lip Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Completed Suicide (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 6 (6)
Depression Suicidal (Psychiatric disorders) | 2 (2)
Major Depression (Psychiatric disorders) | 1 (1)
Mania (Psychiatric disorders) | 2 (2)
Suicidal Ideation (Psychiatric disorders) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone (N=813)
Nausea (Gastrointestinal disorders) | 62 (90)
Akathisia (Nervous system disorders) | 66 (84)
Headache (Nervous system disorders) | 63 (76)
Parkinsonism (Nervous system disorders) | 43 (54)
Anxiety (Psychiatric disorders) | 47 (56)
Insomnia (Psychiatric disorders) | 52 (60)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In addition to the <60-180 day restriction above, since this is a multicenter study, 1st publication of study results shall be made with other participating study sites as a multicenter publication; provided, if a multicenter publication is not forthcoming within 24 months following completion of study at all sites, the PI shall be free to publish.